CLINICAL TRIAL: NCT00211952
Title: A Randomized, Double Blind, Placebo Controlled Phase III Trial Evaluating the Role of Adjuvant Celecoxib in Completely Resected, High-Risk (pN1-2) Non-Small Cell Lung Cancer (NSCLC) Patients
Brief Title: Adjuvant Celecoxib in Completely Resected pN1-2 NSCLC Patients
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Collaborators: Central and Eastern European Oncology Group (Other); Stowarzyszenie Ludzi Wyleczonych z Raka Płuca (Unknown); Pharmacia (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0102 PLCSG
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib

INTERVENTIONS:
Drug: celecoxib

SUMMARY:
The aim of the study is to assess the influence of celecoxib on relapse-free survival in completely resected patients with poor prognosis indicated by metastatic involvement of intrapulmonary/hilar (pN1) or ipsilateral mediastinal (pN2) lymph nodes. Celecoxib, a selective oral COX-2 inhibitor, was found to exert significant anti-proliferative activity against a variety of tumor cell lines in vitro, including NSCLC. COX-2 is frequently up-regulated in NSCLC cell lines and archival tumor samples. Its high expression was also correlated with poor prognosis of the patients. A clinical trial addressing the role of celecoxib as adjuvant treatment in radically operated patients with high risk of relapse is warranted.

DETAILED DESCRIPTION:
1. Rationale and objectives

   To assess the influence of celecoxib on relapse-free survival in completely resected patients with poor prognosis indicated by metastatic involvement of intrapulmonary/hilar (pN1) or ipsilateral mediastinal (pN2) lymph nodes. Celecoxib, a selective oral COX-2 inhibitor, was found to exert significant anti-proliferative activity against a variety of tumor cell lines in vitro, including NSCLC. COX-2 is frequently up-regulated in NSCLC cell lines and archival tumor samples. Its high expression was also correlated with poor prognosis of the patients. Proposed mechanisms of action of selective COX-2 inhibitors include inhibition of angiogenesis, inhibition of matrix metalloproteinase-2 expression and induction of apoptosis. A clinical trial addressing the role of celecoxib as adjuvant treatment in radically operated patients with high risk of relapse is warranted.
2. Study design

   A multicenter, international, randomized, double-blind, placebo controlled phase III clinical trial
3. Primary endpoint

   The primary endpoint will be relapse-free survival (time to local or distant relapse) during the study.
4. Other endpoints

   Secondary end-points will include:
   * overall survival (time to death of any cause)
   * the safety of the long-term administration of celecoxib
5. Statistical methods

   The primary objective, i.e. relapse-free survival (RFS), will be recorded as time from randomization to date of local or distant relapse (date of radiological imaging demonstrating relapse or date of histological confirmation of relapse or date of relapse on clinical examination, if above data are not available) or death of any cause, whichever occurs first. Patients alive without relapse at the end of their follow-up will be considered censored observations.

   The study aims at the verification of the null hypothesis Ho : RFS in the control group = RFS in the treated group vs. the alternative HA : RFS in the control group ≠RFS in the treated group Primary and secondary efficacy analyses will be performed using intention-to-treat principle.

   The distribution of RFS and OS in the compared treatment arms will be summarized graphically using the Kaplan-Meier method and compared by the log-rank test. The result of the test will be assessed using the 5% significance level (two-sided).

   The effect of the treatment on the distribution of RFS and OS will be evaluated by the score test based on the Cox proportional hazards model, which will include stratification and other relevant clinical factors as covariates.

   The proportion of patients experiencing any AE, any serious AE, and specific types of AEs and proportion of withdrawals will be compared between the treatment arms using the chi-square test at the 5% significance level (two-sided).
6. Translational research A research project evaluating immunohistochemical expression of COX-2, VEGF and CD34 as a marker of vascular density will be performed. These parameters will be analyzed in a central laboratory by two independent pathologists involved in angiogenesis research. Immunohistochemical methods will be carefully validated before commencement of translational research part of the study.

   The study centers will be requested to provide post-operative tissue samples (paraffin-embedded blocks or 5 unstained slides) from the primary tumor.
7. Medication

Trt.groups Drug Form Route Dose interval Dosing No. of patients

1. Celecoxib tablets p.o. 400 mg 12 h 271
2. Placebo tablets p.o. 400 mg 12 h 271

ELIGIBILITY:
Eligibility criteria:

* Completely resected (R0), histologically confirmed NSCLC with pathological T1-T3 category and pathological proof of N1 or N2 disease
* Adequate pre-surgical disease assessment (chest CT and upper abdominal CT - mandatory; mediastinoscopy or PET mandatory if clinical N2 is suspected on chest CT; other examinations according to signs and symptoms to exclude metastatic disease)
* Adequate lymph node sampling
* Randomization between 14 and 42 days after surgery
* Adequate post-surgical recovery
* Age > 18 years
* WHO Performance Status 0 or 1
* Adequate liver and renal function (ALT < 1.5 ULN, bilirubin within normal limits, creatinine < 1.5 ULN) and adequate haematology (haemoglobin >11g/dL, WBC>2.000/L, PLT>100.000/L)
* Written informed consent
* No previous treatment with chemotherapy
* No histological diagnosis of SCLC or mixed NSCLC/SCLC type
* No apparent involvement of mediastinal lymph nodes at preoperative staging (cN2)
* No evidence of metastatic disease (M1)
* Stable medical conditions (e.g. no myocardial infarction within 12 months, unstable angina, active psychiatric disorder)
* No active infection
* No history of malignancy other than basal-cell skin cancer or in situ cervical cancer
* No history of severe renal or liver insufficiency
* No history of a recent gastrointestinal bleeding or active ulcer disease or extensive gastro-intestinal surgery that may affect the drug absorption
* No participation in any investigational study within 30 days prior to enrollment
* No pregnancy or lactation or inadequate contraception
* No known hypersensitivity to celecoxib, other COX-2 inhibitors or aspirin (aspirin triad)
* No chronic use of NSAID's (selective inhibitors of COX-2 and non- selective COX inhibitors), acetylsalicylic acid (aspirin) nor oral steroids >14 days during one month prior to surgery nor anticipated chronic use of the above drugs during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542
Dates: Start 2004-03

PRIMARY OUTCOMES:
time to progression

SECONDARY OUTCOMES:
overall survival
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Jassem, Professor, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland